CLINICAL TRIAL: NCT03418584
Title: Application of hybridAPC in the Treatment of Barrett: a Multicenter, Prospective Study
Brief Title: Application of hybridAPC in the Treatment of Barrett
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); The First Affiliated Hospital of Soochow University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHD2017
Record Dates: First submitted 2018-01-10; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Barrett's Esophagus
Keywords: argon plasma coagulation; submucosal injection; Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HybridAPC (Experimental): The patient with Barrett's esophagus is treatment by HybridAPC.
  Interventions: Device: HybridAPC

INTERVENTIONS:
Device: HybridAPC — HybridAPC is a device which combines submucosal fluid injection with APC

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the new technique of HybridAPC in the treatment of Barrett.

DETAILED DESCRIPTION:
After thermal ablation of Barrett's esophagus, stricture formation is reported in 5 to over 10% of patients. Submucosal fluid injection prior to ablation may lower the risk of stricture formation. The new technique of HybridAPC which combines submucosal injection with APC is considered to reduce the complication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age is from 18 to 70.
2. Patients who were diagnosed with Barrett's esophagus.
3. Informed consent.

Exclusion Criteria:

1. Patient with severe cardiopulmonary dysfunction is unable to tolerated by endoscopy.
2. Severe bleeding tendency.
3. Poor compliance.
4. Patient is very ill and life expectancy is less than 2 years.
5. Esophageal varices or venous aneurysms, and no effective prevention or treatment for bleeding.
6. Severe esophageal stenosis.
7. Pregnancy.
8. Lesion is located in esophageal diverticulum or spread their diverticulum.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-12-05 (Actual); Primary Completion 2020-12-05 (Estimated); Study Completion 2021-12-05 (Estimated)

PRIMARY OUTCOMES:
radical rate | 3 months
  Radical rate was defined as it that after 3 months of treatment, the primary lesion area returning to normal is reconfirmed by pathological diagnosis.

SECONDARY OUTCOMES:
recurrence | 3 months
  Recurrence was defined as it that after 3 months of treatment, Barrett's esophagus is reconfirmed by pathological diagnosis in the primary lesion again.
adverse event | 1 year
  Adverse event was defined as any device treatment-related adverse event such as bleeding and perforation
operation time | 1 day
  Operation time was defined as the time from the beginning of submucosal injection to the final end of ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D, Principal Investigator — Changhai Hospital
Locations (1):
- Department of Gastroenterology, Changhai Hospital, Second Military Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fitzgerald RC, di Pietro M, Ragunath K, Ang Y, Kang JY, Watson P, Trudgill N, Patel P, Kaye PV, Sanders S, O'Donovan M, Bird-Lieberman E, Bhandari P, Jankowski JA, Attwood S, Parsons SL, Loft D, Lagergren J, Moayyedi P, Lyratzopoulos G, de Caestecker J; British Society of Gastroenterology. British Society of Gastroenterology guidelines on the diagnosis and management of Barrett's oesophagus. Gut. 2014 Jan;63(1):7-42. doi: 10.1136/gutjnl-2013-305372. Epub 2013 Oct 28. PMID 24165758
- [Result] Manner H, May A, Kouti I, Pech O, Vieth M, Ell C. Efficacy and safety of Hybrid-APC for the ablation of Barrett's esophagus. Surg Endosc. 2016 Apr;30(4):1364-70. doi: 10.1007/s00464-015-4336-1. Epub 2015 Jun 24. PMID 26104794
- [Result] Manner H, Neugebauer A, Scharpf M, Braun K, May A, Ell C, Fend F, Enderle MD. The tissue effect of argon-plasma coagulation with prior submucosal injection (Hybrid-APC) versus standard APC: A randomized ex-vivo study. United European Gastroenterol J. 2014 Oct;2(5):383-90. doi: 10.1177/2050640614544315. PMID 25360316
- [Result] Fujishiro M, Kodashima S, Ono S, Goto O, Yamamichi N, Yahagi N, Kashimura K, Matsuura T, Iguchi M, Oka M, Ichinose M, Omata M. Submucosal Injection of Normal Saline can Prevent Unexpected Deep Thermal Injury of Argon Plasma Coagulation in the in vivo Porcine Stomach. Gut Liver. 2008 Sep;2(2):95-8. doi: 10.5009/gnl.2008.2.2.95. Epub 2008 Sep 30. PMID 20485617
- [Result] Fujishiro M, Yahagi N, Nakamura M, Kakushima N, Kodashima S, Ono S, Kobayashi K, Hashimoto T, Yamamichi N, Tateishi A, Shimizu Y, Oka M, Ichinose M, Omata M. Submucosal injection of normal saline may prevent tissue damage from argon plasma coagulation: an experimental study using resected porcine esophagus, stomach, and colon. Surg Laparosc Endosc Percutan Tech. 2006 Oct;16(5):307-11. doi: 10.1097/01.sle.0000213739.85277.3d. PMID 17057569